CLINICAL TRIAL: NCT02495233
Title: A Phase 1b/2 Study of ASP2215 in Combination With Erlotinib in Subjects With EGFR Activating Mutation-Positive (EGFRm+) Advanced NSCLC Who Have Acquired Resistance to an EGFR Tyrosine Kinase Inhibitor (TKI)
Brief Title: A Study of ASP2215 in Combination With Erlotinib in Subjects With Epidermal Growth Factor Receptor (EGFR) Activating Mutation-Positive (EGFRm+) Advanced Non-Small-Cell Lung Cancer (NSCLC) Who Have Acquired Resistance to an EGFR Tyrosine Kinase Inhibitor (TKI)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study terminated due to adverse events related to the combination therapy
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2215-CL-5101
Record Dates: First submitted 2015-07-08; First posted 2015-07-13 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: Erlotinib; ASP2215; NSCLC; Gilteritinib; Non-Small-Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — gilteritinib; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gilteritinib 120mg + Erlotinib 150mg (Experimental): Gilteritinib was administered in combination with erlotinib orally once daily.
  Interventions: Drug: Gilteritinib; Drug: Erlotinib
- Gilteritinib 80mg+ Erlotinib 150mg (Experimental): Gilteritinib was administered in combination with erlotinib orally once daily.
  Interventions: Drug: Gilteritinib; Drug: Erlotinib

INTERVENTIONS:
Drug: Gilteritinib — oral
Drug: Erlotinib — oral
  Other Names: Tarceva

SUMMARY:
The purpose of the Phase 1b part of the study was to evaluate the safety and tolerability of ASP2215 in combination with erlotinib and determine the recommended phase 2 dose (RP2D) of ASP2215. The purpose of the Phase 2 part of the study was to evaluate the objective response rate (ORR) of the RP2D of ASP2215 in combination with erlotinib.

DETAILED DESCRIPTION:
No patients were enrolled in the Phase 2 part of the study. Phase 2 endpoints were not analyzed.

ELIGIBILITY:
IInclusion Criteria:

* Participant had histologically or cytologically confirmed metastatic or locally advanced, unresectable non-small-cell lung cancer (NSCLC).
* Participant had a documented exon 19 deletion or exon 21 L858R EGFR activating mutation.
* Participant had received prior treatment with any EGFR tyrosine kinase inhibitor
* Participant had Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 2 at screening.
* Participant had adequate organ function.
* Female participant must either:

  * Be of nonchildbearing potential:
  * Or, if of childbearing potential,

    1. Agree not to try to become pregnant during the study and for 45 days after the final study drug administration
    2. And had a negative serum pregnancy test at screening
    3. And, if heterosexually active, agreed to consistently use 2 forms of highly effective birth control
* Male participant and their female spouse/partners who were of childbearing potential must be using highly effective contraception consisting of 2 forms of birth control
* Phase 1b Participants only:

  * Participant was not expected to show a therapeutic response to existing available treatment.
  * Intervening anticancer treatment subsequent to the EGFR TKI was allowed (but not required).
* Additional inclusion criteria for phase 2 Participants only:

  * Participant had a NSCLC tissue sample obtained after participant developed resistance to EGFR TKI therapy that was available for central testing.
  * Participant's baseline tumor specimen (obtained after participant developed resistance to EGFR TKI therapy) is T790M negative.
  * Participant received an EGFR TKI for at least 6 months and progressed on this therapy within the past 28 days.
  * Participant had not had any intervening anticancer treatment subsequent to the EGFR TKI with the exception of radiotherapy which was allowed if it occurred at least 14 days prior to the first dose of study drug.
  * Participant had at least 1 measureable lesion (not including any lesion that was irradiated) based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

Exclusion Criteria:

* Participant had an ongoing toxicity greater than or equal to grade 3 (NCI CTCAE version 4.03) attributable to prior NSCLC treatment at the time of screening.
* Participant received any agent with antitumor activity (other than an EGFR inhibitor, including a T790M inhibitor) including chemotherapy, radiotherapy, immunotherapy, within 14 days prior to the first dose of study drug (palliative radiotherapy is allowed).
* Participant received ASP2215 previously.
* Participant received blood transfusions or hematopoietic growth factor therapy within 14 days prior to the first dose of study drug.
* Participant had a major surgical procedure (other than study-related biopsy) within 14 days prior to the first dose of study drug, or a major surgical procedure was planned to occur during the study.
* Participant had active hepatitis B or C or other active hepatic disorder.
* Participant t was known to have human immunodeficiency virus (HIV) infection.
* Participant had symptomatic central nervous system (CNS) metastasis. Participants with asymptomatic, untreated CNS metastases were allowed. Participants with previously treated and currently asymptomatic CNS metastases were eligible provided they met the following:

  * Any whole brain radiotherapy (WBRT) was completed at least 2 weeks prior to the first dose of study drug.
  * Any stereotactic radiosurgery (SRS) was completed at least 1 week prior to the first dose of study drug.
  * Participant did not require steroids or did not require escalating doses of steroids for at least 2 weeks prior to the first dose of study drug.
* Participant had evidence of active infection requiring systemic therapy within 14 days prior to the first dose of study drug.
* Participant had uncontrolled hypertension.
* Participant had severe or uncontrolled systemic diseases or active bleeding diatheses.
* Participant had history of drug-induced interstitial lung disease or any evidence of active interstitial lung disease.
* Participant had ongoing cardiac arrhythmia (including atrial fibrillation) that was grade ≥ 2.
* Participant currently had Class 3 or 4 New York Heart Association congestive heart failure.
* Participant had history of severe/unstable angina, myocardial infarction or cerebrovascular accident within 6 months prior to the first dose of study drug.
* Participant had history of gastrointestinal ulcer within 28 days prior to the first dose of study drug.
* Participant had a history of gastrointestinal bleeding within 90 days prior to the first dose of study drug.
* Participant had concurrent corneal disorder or any ophthalmologic condition which makes the participant unsuitable for study participation .
* Participant had any condition which made the participant unsuitable for study participation.
* Participant had hypokalemia or hypomagnesemia at screening.
* Participant had QTcF interval > 450 ms on 12-lead ECG at screening.
* Participant was known to have long QT syndrome.
* Participant was taking medication known to prolong the QT interval.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-09-08 (Actual); Primary Completion 2016-09-28 (Actual); Study Completion 2016-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (4):
- Japan (4):
  - Site JP81004, Fukuoka Minami-ku, Fukuoka
  - Site JP81005, Osakasayama, Osaka
  - Site JP81003, Suntogun Nagaizumicho,Shizuoka
  - Site JP81002, Tokyo

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/hcp/study.aspx?ID=286

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with Epidermal growth factor receptor (EGFR) activating mutation-positive (EGFRm+) advanced NSCLC who have acquired resistance to an EGFR Tyrosine kinase inhibitor (TKI) were enrolled in 4 study sites in Japan.
Pre-assignment Details: Eligible participants received gilteritinib in combination with erlotinib 150 mg. At least 3, and no more than 12, dose-limiting toxicity (DLT)-evaluable patients were to be enrolled in a given dose cohort. Dose escalation, cohort expansion or de-escalation decisions were to be guided by a modified toxicity probability interval design.
Period: Overall Study
Arm/Group | Gilteritinib 120mg + Erlotinib 150mg | Gilteritinib 80mg+ Erlotinib 150mg
Started | 3 | 7
Completed | 3 | 6
Not Completed | 0 | 1
Not completed — Miscellaneous | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAF) consisted of all participants who received at least one dose of study drugs.
Groups:
- Total: Total of all reporting groups
Arm/Group | Gilteritinib 120mg + Erlotinib 150mg | Gilteritinib 80mg+ Erlotinib 150mg | Total
Number analyzed (Participants) | 3 | 7 | 10
Age, Continuous [Mean (Standard Deviation); unit: year] | 70.3 (8.4) | 61.4 (5.9) | 64.1 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 1 | 3 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 7 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 7 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Time Frame: Cycle 1 and Cycle ≥2 (up to 141 days)
Population: Safety Analysis Set (SAF) consisted of all participants who received at least one dose of study drugs. DLT evaluable set (DES), was a subset of SAF and included participants who were either administered with at least 75% of planned dose during cycle 1 or experienced DLT during cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Gilteritinib 120mg + Erlotinib 150mg | Gilteritinib 80mg+ Erlotinib 150mg
Number analyzed (Participants) | 3 | 6
Participants
  Cycle 1 | 2 | 2
  Cycle ≥2 | 0 | 1

2. Primary Outcome: Number of Participants With Adverse Events
Description: Treatment-emergent adverse events (TEAE) was defined as an adverse event (AE) that started after administration of the study drugs and occurred within 30 days of the last dose of the study drugs. If a participant experienced an event both during the preinvestigational period and during the investigational period, the event was considered a TEAE only if it worsened in severity.
Time Frame: From first dose of study drug up to 30 days after the last dose of study (maximum study drug exposure 114 days)
Population: SAF
Measure: Count of Participants; unit: Participants
Arm/Group | Gilteritinib 120mg + Erlotinib 150mg | Gilteritinib 80mg+ Erlotinib 150mg
Number analyzed (Participants) | 3 | 7
Participants
  Any TEAEs | 3 | 7
  Drug-related TEAEs | 3 | 7
  TEAEs leading to death | 0 | 0
  Serious TEAEs | 2 | 3
  Drug-related serious TEAEs | 2 | 2
  TEAEs leading to withdrawal of treatment | 2 | 2
  Drug-related TEAEs leading to withdrawal of treat. | 2 | 2

3. Secondary Outcome: Area Under the Concentration-time Curve at 24 Hours (AUC24) for Gilteritinib
Time Frame: 0, 0.5, 1, 2, 4, 6, 24 hours post-dose on Days 1 and 28 of cycle 1
Population: Pharmacokinetic Analysis Set (PKAS) consisted of all participants who received at least 1 dose of study drugs for whom sufficient plasma concentration data were available to facilitate derivation of at least 1 pharmacokinetic parameter and for whom the time of dosing on the day of sampling was known.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Gilteritinib 120mg + Erlotinib 150mg | Gilteritinib 80mg+ Erlotinib 150mg
Number analyzed (Participants) | 3 | 7
h*ng/mL
  Cycle 1 Day 1 | 2950 (1128) | 1885 (685.6)
  Cycle 1 Day 28: number analyzed (Participants) | 1 | 3
  Cycle 1 Day 28 | 12203 (NA) — There was only 1 subject, the mean was the value for that 1 subject. The SD could not be calculated so NA would be entered. | 8342 (3023)

4. Secondary Outcome: Maximum Concentration (Cmax) for Gilteritinib
Time Frame: 0, 0.5, 1, 2, 4, 6, 24 hours post-dose on Days 1 and 28 of cycle 1
Population: PKAS
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Gilteritinib 120mg + Erlotinib 150mg | Gilteritinib 80mg+ Erlotinib 150mg
Number analyzed (Participants) | 3 | 7
ng/mL
  Cycle 1 Day 1 | 210.3 (107.4) | 119 (47.65)
  Cycle 1 Day 28: number analyzed (Participants) | 1 | 3
  Cycle 1 Day 28 | 637 (NA) — There was only 1 subject, the mean was the value for that 1 subject. The SD could not be calculated so NA would be entered. | 408.3 (136.6)

5. Secondary Outcome: Time After Dosing When Cmax Occurs (Tmax) for Gilteritinib
Time Frame: 0, 0.5, 1, 2, 4, 6, 24 hours post-dose on Days 1 and 28 of cycle 1
Population: PKAS
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Gilteritinib 120mg + Erlotinib 150mg | Gilteritinib 80mg+ Erlotinib 150mg
Number analyzed (Participants) | 3 | 7
hr
  Cycle 1 Day 1, | 3.961 (0.08221) | 3.762 (0.8109)
  Cycle 1 Day 28: number analyzed (Participants) | 1 | 3
  Cycle 1 Day 28 | 2.00 (NA) — There was only 1 subject, the mean was the value for that 1 subject. The SD could not be calculated so NA would be entered. | 4.594 (1.044)

6. Secondary Outcome: Concentration Immediately Prior to Dosing at Multiple Dosing (Ctrough) of Gilteritinib
Description: All participants in Gilteritinib 120 mg + Erlotinib 150 mg group discontinued before cycle 3.
Time Frame: Predose on Day 1, 3, 8, 15, 22, 28 of cycle 1, Day 1 of cycle 3 and Day 1 of cycle 4
Population: PKAS
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Gilteritinib 120mg + Erlotinib 150mg | Gilteritinib 80mg+ Erlotinib 150mg
Number analyzed (Participants) | 3 | 7
ng/mL
  Predose on Day 1 of cycle 1 | 0 (0) | 0 (0)
  Predose on Day 3 of cycle 1: number analyzed (Participants) | 3 | 6
  Predose on Day 3 of cycle 1 | 112 (21.7) | 110.2 (46.51)
  Predose on Day 8 of cycle 1 | 261.3 (31.66) | 282.9 (136.7)
  Predose on Day 15 of cycle 1: number analyzed (Participants) | 3 | 6
  Predose on Day 15 of cycle 1 | 491.7 (430.5) | 397 (208.9)
  Predose on Day 22 of cycle 1: number analyzed (Participants) | 3 | 6
  Predose on Day 22 of cycle 1 | 466.3 (128.2) | 414.8 (186.1)
  Predose on Day 28 of cycle 1: number analyzed (Participants) | 1 | 4
  Predose on Day 28 of cycle 1 | 430 (NA) — There was only 1 subject, the mean was the value for that 1 subject. The SD could not be calculated so NA would be entered. | 241.3 (114.4)
  Predose on Day 1 of cycle 3: number analyzed (Participants) | 0 | 2
  Predose on Day 1 of cycle 3 |  | 161 (38.18)
  Predose on Day 1 of cycle 4: number analyzed (Participants) | 0 | 2
  Predose on Day 1 of cycle 4 |  | 236 (104.7)

7. Secondary Outcome: AUC24 of Erlotinib
Time Frame: 0, 0.5, 1, 2, 4, 6, 24 hours post-dose on Day 28 of cycle 1
Population: PKAS
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Gilteritinib 120mg + Erlotinib 150mg | Gilteritinib 80mg+ Erlotinib 150mg
Number analyzed (Participants) | 1 | 3
h*ng/mL | 34580 (NA) — There was only 1 subject, the mean was the value for that 1 subject. The SD could not be calculated so NA would be entered. | 54055 (22962)

8. Secondary Outcome: Cmax of Erlotinib
Time Frame: 0, 0.5, 1, 2, 4, 6, 24 hours post-dose on Day 28 of cycle 1
Population: PKAS
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Gilteritinib 120mg + Erlotinib 150mg | Gilteritinib 80mg+ Erlotinib 150mg
Number analyzed (Participants) | 1 | 3
ng/mL | 3050 (NA) — There was only 1 subject, the mean was the value for that 1 subject. The SD could not be calculated so NA would be entered. | 3160 (314.3)

9. Secondary Outcome: Tmax of Erlotinib
Time Frame: 0, 0.5, 1, 2, 4, 6, 24 hours post-dose on Day 28 of cycle 1
Population: PKAS
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Gilteritinib 120mg + Erlotinib 150mg | Gilteritinib 80mg+ Erlotinib 150mg
Number analyzed (Participants) | 1 | 3
hr | 2.00 (NA) — There was only 1 subject, the mean was the value for that 1 subject. The SD could not be calculated so NA would be entered. | 2.633 (1.185)

10. Secondary Outcome: Ctrough of Erlotinib
Time Frame: Day 8, 15, 22, 28 of cycle 1
Population: PKAS
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Gilteritinib 120mg + Erlotinib 150mg | Gilteritinib 80mg+ Erlotinib 150mg
Number analyzed (Participants) | 3 | 7
ng/mL
  Predose of Day 8 of cycle 1 | 1004 (758.7) | 1827 (1392)
  Predose of Day 15 of cycle 1: number analyzed (Participants) | 3 | 6
  Predose of Day 15 of cycle 1 | 1427 (1596) | 2098 (1637)
  Predose of Day 22 of cycle 1: number analyzed (Participants) | 3 | 6
  Predose of Day 22 of cycle 1 | 942.7 (116) | 1999 (1285)
  Predose of Day 28 of cycle 1: number analyzed (Participants) | 1 | 4
  Predose of Day 28 of cycle 1 | 909 (NA) — There was only 1 subject, the mean was the value for that 1 subject. The SD could not be calculated so NA would be entered. | 1368 (1255)

11. Secondary Outcome: Objective Response Rate (ORR) in Phase 1b
Description: ORR was defined as Objective Response Rate (ORR) was the proportion of patients whose best overall response was complete response (CR) or partial response (PR) per RECIST version 1.1. Only patients with measurable disease at baseline were to be included in the analysis of ORR.
Time Frame: End of treatment (approximately 4 months)
Population: ASAT consisted of all participants allocated to treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Gilteritinib 120mg + Erlotinib 150mg | Gilteritinib 80mg+ Erlotinib 150mg
Number analyzed (Participants) | 3 | 6
percentage of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days after the last dose of study (maximum study drug exposure 114 days)
Description: Safety Analysis Set (SAF) consisted of all participants who received at least one dose of study drugs.
Arm/Group | Gilteritinib 120mg + Erlotinib 150mg | Gilteritinib 80mg+ Erlotinib 150mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/7
Serious Adverse Events (participants affected / at risk) | 2/3 | 3/7
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gilteritinib 120mg + Erlotinib 150mg (N=3) | Gilteritinib 80mg+ Erlotinib 150mg (N=7)
Alanine aminotransferase increased (Investigations) | 2 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gilteritinib 120mg + Erlotinib 150mg (N=3) | Gilteritinib 80mg+ Erlotinib 150mg (N=7)
Diarrhoea (Gastrointestinal disorders) | 3 | 4
Constipation (Gastrointestinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastric disorder (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 4
Aspartate aminotransferase increased (Investigations) | 1 | 5
Blood creatine phosphokinase increased (Investigations) | 2 | 3
Blood alkaline phosphatase increased (Investigations) | 0 | 3
Blood creatinine increased (Investigations) | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 2
Aldolase increased (Investigations) | 0 | 1
Amylase increased (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Myoglobin blood increased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 2 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Paronychia (Infections and infestations) | 1 | 2
Acne pustular (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Gastroenteritis staphylococcal (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2
Dysgeusia (Nervous system disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Malaise (General disorders) | 2 | 0
Fatigue (General disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 2
Proteinuria (Renal and urinary disorders) | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.